CLINICAL TRIAL: NCT00515463
Title: A Multi-Center, Randomized, Open-Label Study to Assess the Immunogenicity and Safety of Denosumab in Pre-filled Syringe Compared to Vial in Subjects With Low Bone Mineral Density
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060237
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2013-10-31 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-08

CONDITIONS: Low Bone Mineral Density; Osteopenia; Osteoporosis
Keywords: Osteopenia; Osteoporosis; AMG 162; Postmenopausal; Pre-filled syringe
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Denosumab

ARMS (2):
- Denosumab - Vial (Experimental): Participants received denosumab 60 mg subcutaneous injection using a standard vial on Day 1 and at Month 6.
  Interventions: Biological: denosumab
- Denosumab - Prefilled syringe (Experimental): Participants received denosumab 60 mg subcutaneous injection using a pre-filled syringe on Day 1 and at Month 6.
  Interventions: Biological: denosumab

INTERVENTIONS:
Biological: denosumab — 60 mg denosumab in 1mL
  Arms: Denosumab - Vial
Biological: denosumab — 60 mg denosumab in 1mL
  Arms: Denosumab - Prefilled syringe

SUMMARY:
The purpose of this study is to compare the immunogenicity profiles of denosumab pre-filled syringe (PFS) and vial at 6 months in postmenopausal women with low bone mineral density (BMD).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have successfully completed the 20050141 study (NCT00330460):

  * Must have received all SC investigational product administrations in 20050141
  * Must not have taken any proscribed therapies in 20050141
  * Subjects who were in the alendronate or denosumab treatment group are allowed
* Provide signed informed consent before any study-specific procedures are conducted

Exclusion Criteria:

* Any disorder that, in the opinion of the investigator, may compromise the ability of the patient to give written informed consent and/or comply with study procedures including:

  * Any physical or psychiatric disorder
  * Or evidence of alcohol or substance abuse in the last 12 months
* Any clinical evidence, in the medical judgement of the investigator, of the following medical conditions:

  * Impaired thyroid function (subsequent to treatment)
  * Impaired hepatic function
  * Impaired renal function
  * Rheumatoid Arthritis, Paget's disease, Cushing's disease, hyperprolactinemia, or cirrhosis of the liver
  * Known to have tested positive for human immunodeficiency virus, hepatitis C virus, or hepatitis B surface antigen
  * Any metabolic bone disease, eg, osteomalacia or osteogenesis imperfecta, which may interfere with the interpretation of the findings

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who successfully completed Study 20050141 (NCT00330460) were eligible to participate in this study.
  First Subject Enrolled: 30-May-2007 Last Subject Enrolled: 10-Sep-2007
Groups:
- Denosumab - Pre-filled Syringe: Participants received denosumab 60 mg subcutaneous injection using a pre-filled syringe on Day 1 and at Month 6.
Period: Overall Study
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Started | 155 | 156
Received Study Medication | 154 | 156
Completed | 141 | 142
Not Completed | 14 | 14
Not completed — Physician Decision | 4 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 6 | 5
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe | Total
Number analyzed (Participants) | 155 | 156 | 311
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (8.5) | 62.9 (8.9) | 62.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 156 | 311
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 124 | 131 | 255
  Black or African American | 4 | 1 | 5
  Hispanic or Latino | 24 | 18 | 42
  Asian | 3 | 3 | 6
  Japanese | 0 | 2 | 2
  American Indian or Alaska Native | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Tested Positive for Anti-denosumab Antibodies at Month 6
Description: An electrochemiluminescent bridging immunoassay was used to test blood samples for binding antibodies to denosumab.
Time Frame: 6 months
Population: Patients who received ≥ 1 dose of investigational product, have a baseline and ≥ 1 post-baseline antibody assessment and did not have binding anti-denosumab antibodies present at baseline, and with evaluable antibody results at 6 months.
Measure: Number; unit: Participants
Groups:
- Denosumab - Pre-filled Syringe: Participants received denosumab 60 mg subcutaneous injection using a pre-filled syringe (PFS) on Day 1 and at Month 6.
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 146
Participants | 0 | 0
Statistical Analysis 1: Comparison: Denosumab - Vial vs Denosumab - Pre-filled Syringe; Test type: Superiority or Other; Risk Difference (RD) = 0, 95% CI [-0.7 to 0.7] — Risk difference > 0 indicates that incidence of binding anti-denosumab antibodies in denosumab PFS is greater than denosumab vial. 95% CI based on a normal approximation with continuity correction

2. Secondary Outcome: Number of Participants Who Tested Positive for Anti-denosumab Antibodies at Month 12
Description: An electrochemiluminescent bridging immunoassay was used to test blood samples for binding antibodies to denosumab.
Time Frame: 12 months
Population: Patients who received ≥ 1 dose of investigational product, have a baseline and ≥ 1 post-baseline antibody assessment and did not have binding anti-denosumab antibodies present at baseline, and with evaluable antibody results at 12 months.
Measure: Number; unit: Participants
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 140
Participants | 0 | 0
Statistical Analysis 1: Comparison: Denosumab - Vial vs Denosumab - Pre-filled Syringe; Test type: Superiority or Other; Risk Difference (RD) = 0, 95% CI [-0.7 to 0.7]

3. Secondary Outcome: Number of Participants With Neutralizing Antibodies Against Denosumab at Month 12
Description: Samples demonstrating reactivity for binding antibodies to denosumab were to be tested for neutralizing or inhibitory effects in a cell-based bioassay.
Time Frame: Month 12
Population: Patients testing positive for binding antibodies to denosumab.
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Sodium Change From Baseline at Month 1
Description: Laboratory chemistry sodium
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
mmol/L | -0.1 (2.0) | 0.1 (1.7)

5. Secondary Outcome: Sodium Change From Baseline at Month 6
Description: Laboratory chemistry sodium
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
mmol/L | -1.2 (2.0) | -0.9 (1.8)

6. Secondary Outcome: Sodium Change From Baseline at Month 12
Description: Sodium Change From Baseline at Month 12
Time Frame: Baseline, Month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
mmol/L | -0.9 (2.1) | -0.6 (2.0)

7. Secondary Outcome: Potassium Change From Baseline at Month 1
Description: Laboratory chemistry potassium
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
mmol/L | 0.02 (0.37) | 0 (0.39)

8. Secondary Outcome: Potassium Change From Baseline at Month 6
Description: Laboratory chemistry potassium
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
mmol/L | 0.01 (0.43) | -0.07 (0.40)

9. Secondary Outcome: Potassium Change From Baseline at Month 12
Description: Laboratory chemistry potassium
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
mmol/L | 0.07 (0.40) | 0.04 (0.40)

10. Secondary Outcome: Chloride Change From Baseline at Month 1
Description: Laboratory chemistry chloride
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
mmol/L | -0.1 (2.1) | 0.2 (1.9)

11. Secondary Outcome: Chloride Change From Baseline at Month 6
Description: Laboratory chemistry chloride
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
mmol/L | -0.9 (2.3) | -0.4 (2.0)

12. Secondary Outcome: Chloride Change From Baseline at Month 12
Description: Laboratory chemistry chloride
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
mmol/L | -0.2 (2.1) | 0 (2.5)

13. Secondary Outcome: Bicarbonate Change From Baseline at Month 1
Description: Laboratory chemistry bicarbonate
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 145 | 149
mmol/L | -0.3 (2.9) | 0 (2.9)

14. Secondary Outcome: Bicarbonate Change From Baseline at Month 6
Description: Laboratory chemistry bicarbonate
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 141 | 143
mmol/L | 0.2 (2.7) | 0.1 (2.9)

15. Secondary Outcome: Bicarbonate Change From Baseline at Month 12
Description: Laboratory chemistry bicarbonate
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 138 | 139
mmol/L | -0.6 (2.8) | -0.1 (2.8)

16. Secondary Outcome: Magnesium Change From Baseline at Month 1
Description: Laboratory chemistry magnesium
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
mmol/L | 0.001 (0.092) | -0.010 (0.080)

17. Secondary Outcome: Magnesium Change From Baseline at Month 6
Description: Laboratory chemistry magnesium
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
mmol/L | -0.053 (0.073) | -0.064 (0.080)

18. Secondary Outcome: Magnesium Change From Baseline at Month 12
Description: Laboratory chemistry magnesium
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
mmol/L | -0.053 (0.062) | -0.055 (0.074)

19. Secondary Outcome: Blood Urea Nitrogen Change From Baseline at Month 1
Description: Laboratory chemistry blood urea nitrogen
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
mmol/L | 0.01 (1.30) | -0.04 (1.38)

20. Secondary Outcome: Blood Urea Nitrogen Change From Baseline at Month 6
Description: Laboratory chemistry blood urea nitrogen
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
mmol/L | 0.09 (1.40) | 0.11 (1.49)

21. Secondary Outcome: Blood Urea Nitrogen Change From Baseline at Month 12
Description: Laboratory chemistry blood urea nitrogen
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
mmol/L | 0.27 (1.44) | -0.02 (1.50)

22. Secondary Outcome: Creatinine Change From Baseline at Month 1
Description: Laboratory chemistry creatinine
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
umol/L | 0.24 (8.01) | 0.12 (7.76)

23. Secondary Outcome: Creatinine Change From Baseline at Month 6
Description: Laboratory chemistry creatinine
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
umol/L | -0.19 (8.52) | -1.29 (8.23)

24. Secondary Outcome: Creatinine Change From Baseline at Month 12
Description: Laboratory chemistry creatinine
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
umol/L | 1.40 (9.53) | 0.76 (8.28)

25. Secondary Outcome: Aspartate Amino Transferase Change From Baseline at Month 1
Description: Laboratory chemistry aspartate amino transferase
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 146 | 149
U/L | -1.6 (13.0) | 0.4 (4.7)

26. Secondary Outcome: Aspartate Amino Transferase Change From Baseline at Month 6
Description: Laboratory chemistry aspartate amino transferase
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 141 | 144
U/L | -1.6 (13.9) | 0.9 (7.7)

27. Secondary Outcome: Aspartate Amino Transferase Change From Baseline at Month 12
Description: Laboratory chemistry aspartate amino transferase
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 138 | 139
U/L | -1.9 (13.5) | 0.2 (3.9)

28. Secondary Outcome: Alanine Amino Transferase Change From Baseline at Month 1
Description: Laboratory chemistry alanine amino transferase
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 145 | 149
U/L | -3.1 (25.7) | 0.5 (5.5)

29. Secondary Outcome: Alanine Amino Transferase Change From Baseline at Month 6
Description: Laboratory chemistry alanine amino transferase
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 141 | 143
U/L | -1.4 (27.8) | 4.2 (15.2)

30. Secondary Outcome: Alanine Amino Transferase Change From Baseline at Month 12
Description: Laboratory chemistry alanine amino transferase
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 138 | 139
U/L | -2.7 (28.8) | 1.5 (6.3)

31. Secondary Outcome: Total Bilirubin Change From Baseline at Month 1
Description: Laboratory chemistry total bilirubin
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 146 | 149
umol/L | -0.35 (2.53) | -0.02 (2.47)

32. Secondary Outcome: Total Bilirubin Change From Baseline at Month 6
Description: Laboratory chemistry total bilirubin
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 141 | 143
umol/L | -0.30 (2.54) | -0.20 (2.67)

33. Secondary Outcome: Total Bilirubin Change From Baseline at Month 12
Description: Laboratory chemistry total bilirubin
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 138 | 139
umol/L | 0.16 (2.68) | 0.64 (2.74)

34. Secondary Outcome: Albumin Change From Baseline at Month 1
Description: Laboratory chemistry albumin
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
g/L | -0.46 (1.68) | -0.40 (2.05)

35. Secondary Outcome: Albumin Change From Baseline at Month 6
Description: Laboratory chemistry albumin
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
g/L | -0.34 (1.92) | -0.51 (2.19)

36. Secondary Outcome: Albumin Change From Baseline at Month 12
Description: Laboratory chemistry albumin
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
g/L | -0.26 (1.82) | 0 (2.03)

37. Secondary Outcome: Total Protein Change From Baseline at Month 1
Description: Laboratory chemistry total protein
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
g/L | -0.59 (2.67) | -0.54 (3.45)

38. Secondary Outcome: Total Protein Change From Baseline at Month 6
Description: Laboratory chemistry total protein
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
g/L | -0.58 (3.00) | -0.80 (3.33)

39. Secondary Outcome: Total Protein Change From Baseline at Month 12
Description: Laboratory chemistry total protein
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
g/L | -1.35 (2.84) | -0.91 (3.28)

40. Secondary Outcome: Glucose Change From Baseline at Month 1
Description: Laboratory chemistry glucose
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 147 | 149
mmol/L | -0.08 (1.27) | 0.03 (0.69)

41. Secondary Outcome: Glucose Change From Baseline at Month 6
Description: Laboratory chemistry glucose
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 142 | 144
mmol/L | -0.08 (1.37) | 0.05 (0.80)

42. Secondary Outcome: Glucose Change From Baseline at Month 12
Description: Laboratory chemistry glucose
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 139 | 139
mmol/L | -0.06 (1.27) | 0.08 (0.92)

43. Secondary Outcome: Red Blood Cells Change From Baseline at Month 1
Description: Laboratory hematology red blood cells
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^12/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^12/L | 0 (0.21) | 0.02 (0.23)

44. Secondary Outcome: Red Blood Cells Change From Baseline at Month 6
Description: Laboratory hematology red blood cells
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^12/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 142
10^12/L | 0.04 (0.22) | 0.04 (0.22)

45. Secondary Outcome: Red Blood Cells Change From Baseline at Month 12
Description: Laboratory hematology red blood cells
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^12/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 137 | 140
10^12/L | -0.01 (0.22) | 0.02 (0.23)

46. Secondary Outcome: Hemoglobin Change From Baseline at Month 1
Description: Laboratory hematology hemoglobin
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
g/L | -0.97 (6.00) | -0.42 (6.24)

47. Secondary Outcome: Hemoglobin Change From Baseline at Month 6
Description: Laboratory hematology hemoglobin
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 142
g/L | 0.84 (5.83) | 0.96 (6.34)

48. Secondary Outcome: Hemoglobin Change From Baseline at Month 12
Description: Laboratory hematology hemoglobin
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 137 | 140
g/L | -1.74 (6.09) | -0.22 (6.62)

49. Secondary Outcome: Reticulocytes Change From Baseline at Month 1
Description: Laboratory hematology reticulocytes
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^9/L | 3.70 (17.68) | 1.69 (17.41)

50. Secondary Outcome: Reticulocytes Change From Baseline at Month 6
Description: Laboratory hematology reticulocytes
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 142
10^9/L | 19.54 (19.22) | 15.21 (20.69)

51. Secondary Outcome: Reticulocytes Change From Baseline at Month 12
Description: Laboratory hematology reticulocytes
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 137 | 140
10^9/L | 19.09 (19.82) | 15.08 (19.73)

52. Secondary Outcome: Platelets Change From Baseline at Month 1
Description: Laboratory hematology platelets
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 138 | 147
10^9/L | 5.24 (33.20) | 2.48 (36.20)

53. Secondary Outcome: Platelets Change From Baseline at Month 6
Description: Laboratory hematology platelets
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 136 | 142
10^9/L | 28.26 (32.16) | 21.49 (53.82)

54. Secondary Outcome: Platelets Change From Baseline at Month 12
Description: Laboratory hematology platelets
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 133 | 139
10^9/L | 25.19 (42.07) | 15.60 (41.82)

55. Secondary Outcome: White Blood Cells Change From Baseline at Month 1
Description: Laboratory hematology white blood cells
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^9/L | 0.23 (1.07) | 0.01 (1.26)

56. Secondary Outcome: White Blood Cells Change From Baseline at Month 6
Description: Laboratory hematology white blood cells
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 142
10^9/L | 0.22 (1.38) | -0.08 (1.47)

57. Secondary Outcome: White Blood Cells Change From Baseline at Month 12
Description: Laboratory hematology white blood cells
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 137 | 140
10^9/L | 0.47 (1.38) | 0.24 (1.47)

58. Secondary Outcome: Total Neutrophils Change From Baseline at Month 1
Description: Laboratory hematology total neutrophils
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^9/L | 0.11 (0.85) | -0.03 (1.10)

59. Secondary Outcome: Total Neutrophils Change From Baseline at Month 6
Description: Laboratory hematology total neutrophils
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 142
10^9/L | 0.21 (1.23) | -0.02 (1.23)

60. Secondary Outcome: Total Neutrophils Change From Baseline at Month 12
Description: Laboratory hematology total neutrophils
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 136 | 140
10^9/L | 0.38 (1.15) | 0.12 (1.18)

61. Secondary Outcome: Eosinophils Change From Baseline at Month 1
Description: Laboratory hematology eosinophils
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^9/L | -0.002 (0.065) | -0.010 (0.059)

62. Secondary Outcome: Eosinophils Change From Baseline at Month 6
Description: Laboratory hematology eosinophils
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 142
10^9/L | 0.020 (0.075) | 0.013 (0.104)

63. Secondary Outcome: Eosinophils Change From Baseline at Month 12
Description: Laboratory hematology eosinophils
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 136 | 140
10^9/L | -0.008 (0.071) | 0.025 (0.436)

64. Secondary Outcome: Basophils Change From Baseline at Month 1
Description: Laboratory hematology basophils
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^9/L | 0.001 (0.025) | 0 (0.022)

65. Secondary Outcome: Basophils Change From Baseline at Month 6
Description: Laboratory hematology basophils
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 142
10^9/L | 0.012 (0.026) | 0.012 (0.028)

66. Secondary Outcome: Basophils Change From Baseline at Month 12
Description: Laboratory hematology basophils
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 136 | 140
10^9/L | 0.003 (0.026) | 0.006 (0.024)

67. Secondary Outcome: Lymphocytes Change From Baseline at Month 1
Description: Laboratory hematology lymphocytes
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^9/L | 0.12 (0.43) | 0.04 (0.40)

68. Secondary Outcome: Lymphocytes Change From Baseline at Month 6
Description: Laboratory hematology lymphocytes
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^9/L | 0.01 (0.37) | -0.06 (0.45)

69. Secondary Outcome: Lymphocytes Change From Baseline at Month 12
Description: Laboratory hematology lymphocytes
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 136 | 140
10^9/L | 0.08 (0.41) | 0.06 (0.36)

70. Secondary Outcome: Monocytes Change From Baseline at Month 1
Description: Laboratory hematology monocytes
Time Frame: Baseline, month 1
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 1.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 143 | 147
10^9/L | 0 (0.12) | 0.01 (0.11)

71. Secondary Outcome: Monocytes Change From Baseline at Month 6
Description: Laboratory hematology monocytes
Time Frame: Baseline, month 6
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 6.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 140 | 142
10^9/L | -0.03 (0.14) | -0.03 (0.10)

72. Secondary Outcome: Monocytes Change From Baseline at Month 12
Description: Laboratory hematology monocytes
Time Frame: Baseline, month 12
Population: Subjects who received ≥ 1 dose of investigational product with non-missing baseline and non-missing month 12.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 136 | 140
10^9/L | 0.01 (0.13) | 0.03 (0.14)

73. Secondary Outcome: Number of Participants With Laboratory Toxicity CTCAE Grade Greater or Equal to 3
Description: Participants with laboratory toxicity grade 3 (severe) or 4 (life-threatening), based on the Common Terminology Criteria for Adverse Events (CTCAE), version 3.0.
Time Frame: Day 1 to Month 12
Population: Patients who received ≥ 1 dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Number analyzed (Participants) | 154 | 156
Participants
  Number of patients with CTCAE grade 3 or 4 | 2 | 2
  Sodium - Grade 3 below normal (< 130 - 120 mmol/L) | 0 | 1
  Potassium - Grade 3 above normal (>6.0-7.0 mmol/L) | 0 | 1
  Magnesium -Grade 3 above normal (>1.23-3.30mmol/L) | 2 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Denosumab - Vial | Denosumab - Pre-filled Syringe
Serious Adverse Events (participants affected / at risk) | 7/154 | 12/156
Other Adverse Events (participants affected / at risk) | 32/154 | 49/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab - Vial (N=154) | Denosumab - Pre-filled Syringe (N=156)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab - Vial (N=154) | Denosumab - Pre-filled Syringe (N=156)
Sinusitis (Infections and infestations) | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 5 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 11
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.